CLINICAL TRIAL: NCT05406804
Title: The Influence of Olfactory Stimulation of Breast Milk on the Stability of Physiological Indicators of Very Low Birth Weight Infants
Brief Title: Olfactory Stimulation for Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NICU olfactory stimulation-01
Record Dates: First submitted 2022-02-14; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-04

CONDITIONS: Very Low Birth Weight Infant
Keywords: Olfactory stimulation; Heart rate; Oxygen saturation; Respiratory rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast milk olfactory stimulation care (Experimental): Let premature babies smell their mother's breast milk
  Interventions: Behavioral: Olfactory stimulation
- Routine care (Active Comparator): Prevent premature babies from smelling their mother's breast milk
  Interventions: Behavioral: Routine nursing care

INTERVENTIONS:
Behavioral: Olfactory stimulation — 1) For the premature infants who use non-invasive ventilation, place a single layer of gauze soaked in breast milk on the air outlet of the non-invasive ventilator. When inhaling oxygen with a high-flow nasal cannula, the same measure is performed, and the breast milk and sterile gauze soaked in breast milk are replaced every 4 hours. 2) For the premature infants who withdrawn from assisted ventilation, place the breast pad near the infants' nose, and replace the breast milk pad every 4 hours. Acquisition of breast milk pads: use the same brand of breast milk pads; put the breast milk pads used between 00:00 and 07:00 every day (use time > 2 hours) into the same brand of milk storage bags, and use two left and right at the same time. 3) If the premature infants don't have any ventilation support, the breast milk stimulation method is the same as 2). This intervention will continue until premature infants discharge from hospital.
  Arms: Breast milk olfactory stimulation care
Behavioral: Routine nursing care — Nursing is performed according to existing nursing practices. Nasal feeding is generally used.
  Arms: Routine care

SUMMARY:
This is a RCT study examining whether odor administration to mothers of very low birth weight infants promotes stabilization of vital signs compared with common nursing care. This study used breast milk olfactory stimuli familiar and liked by premature infants to understand the effects of olfactory stimuli on the physiological indicators of very low birth weight infants, the effect on the time of complete enteral nutrition, and the effects on growth and development of very low birth weight infants.

DETAILED DESCRIPTION:
Fluctuations in vital signs of very low birth weight infants may lead to poor prognosis. Research Objectives:

To evaluate the effect of olfactory stimulation of breast milk on the stability of physiological indexes of very low birth weight infants Subjects: Very low birth weight infants whose gestational age are less than 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth <32 weeks;
* Birth weight < 1500 g;
* Admission to hospital within 24 hours after birth;
* Mother can provide breast milk

Exclusion Criteria:

* Severe congenital malformations;
* Complicated congenital heart disease;
* Congenital gastrointestinal disease;
* Intraventricular hemorrhage

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Ratio of stable heart rate | During the procedure.
  During the intervention period, the frequency of the measured heart rate between 120 bpm and 160bpm divide the total frequency of heart rate monitoring. The heart rate, blood oxygen saturation and other data will be automatically uploaded to the system by the electrocardiogram monitor every minute, one for each one every minute, which is downloaded by the researcher and then entered into the computer.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu L, Tao Y, Jia P, Li L, Lv T, Wang L, Song Q, Huan X, Liu C, Dou Y, Xuan Y, Hu XJ. Effect of breast milk olfactory experience on physiological indicators in very low birth weight infants: a randomized clinical trial. Sci Rep. 2025 Jul 1;15(1):20590. doi: 10.1038/s41598-025-05809-0. PMID 40596001